CLINICAL TRIAL: NCT02910869
Title: PREDICT: Nutrigenetic Profile of Patients With Weight Loss Success in MOVE! and TeleMOVE! Programs
Brief Title: PREDICT: Nutrigenetic Profile of Patients With Weight Loss Success
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Pathway Genomics Corp (Unknown)
Responsible Party: Principal Investigator, Amir Zarrinpar, MD, San Diego Veterans Healthcare System
Other Study IDs: H150148
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Successful weight loss: Patients who have lost =>5% of their weight after completing MOVE! or TeleMOVE!
  Interventions: Genetic: Pathway Genomics FIT test
- Unsuccessful weight loss: Patients who have lost <5% of their weight after completing MOVE! or TeleMOVE!
  Interventions: Genetic: Pathway Genomics FIT test

INTERVENTIONS:
Genetic: Pathway Genomics FIT test

SUMMARY:
This observational study will investigate the potential clinical utility of the Pathway Fit® test by investigating whether patients who successfully lose weight (defined as losing at least 5% of body weight 8 weeks after initiation) in the MOVE! or TeleMOVE! Weight Management programs have a distinct nutrigenetic profile over those that were unable to lose a significant amount of weight. We will use electronic records to identify all individuals who have successfully completed the MOVE! program (i.e. attended the full 8 week course) or TeleMOVE! program. In addition we will find age- and gender- matched individuals who attended and completed the MOVE! or TeleMOVE! programs but did not lose weight. After completion of the MOVE! or TeleMOVE! programs Veterans will submit a saliva sample for the Pathway Fit® test. Also, blood will be collected for storage for further studies on metabolomics. The start and end weight of all participants will be recorded. The nutrigenic profiles of those with successful weight loss will be compared to those less successful to determine if this cohort has a particular genetic profile.

DETAILED DESCRIPTION:
The overall prevalence of metabolic syndrome in the general US population is estimated to be 22-34.5% with greater prevalence in certain populations (e.g. Mexican and African Americans, women). These numbers have been consistent with the rise of prevalence of obesity in the US population to 34.9%, which has remained stable over the last 10 years. Veterans are particularly predisposed to metabolic syndrome since the prevalence of obesity is much higher among their ranks. Since the annual medical cost of those who are obese or have metabolic syndrome is $1429 higher than those at a healthy weight, the impact on the cost of healthcare for Veterans can be potentially tremendous. This is mainly since obesity is strongly associated with many chronic diseases, including type 2 diabetes, cardiovascular disease, some types of cancer (endometrial, postmenopausal breast, kidney, and colon), musculoskeletal disorders, sleep apnea, and gallbladder disease.

In order to combat the obesity epidemic in Veterans, the U.S. Department of Veterans Affairs created the MOVE! Weight Management Program (MOVE!) in 2006. MOVE! is an evidence-based weight-management program designed for patients followed in primary care clinics and who have a BMI of ≥30kg/m2 or with a BMI of ≥25kg/m2 with 1 or more obesity-related conditions (e.g. diabetes, hypertension, dyslipidemia). The efficacy of the program is measured by the % of patients who losing at least 5% of body weight at 8 weeks and 6 months after first session. In addition, TeleMOVE! is a program recently initiated within the VA system to help individuals who cannot make it to the VA MOVE! program due to their work schedule or distance from VA clinic.

This observational study will investigate the potential clinical utility of the Pathway Fit® test by investigating whether patients who successfully lose weight (defined as losing at least 5% of body weight 8 weeks after initiation) in the MOVE! or TeleMOVE! programs have a distinct nutrigenetic profile over those that were unable to lose a significant amount of weight. We will use electronic records to identify all individuals who have successfully completed the MOVE! program (i.e. attended the full 8 week course) or TeleMOVE! program. In addition we will find age- and gender- matched individuals who attended and completed the MOVE! Or TeleMOVE! programs but did not lose weight. After completion of the MOVE! Or TeleMOVE! programs Veterans will submit a saliva sample for the Pathway Fit® test. The start and end weight of all participants will be recorded. The nutrigenic profiles of those with successful weight loss will be compared to those less successful to determine if this cohort has a particular genetic profile. Also, blood will be collected for storage for further studies on metabolomics.

To encourage participation, participants will be reimbursed for their participation in the study and the Pathway Fit® test results will be provided to all. Comparisons on all pertinent measures will be made between those achieving at least 5% weight loss and those that did not.

Upon completion of the study, the clinical utility of the Pathway Fit® test can be further investigated to determine if the successful nutrigenic profile can predict clinical outcomes of the participants in the MOVE! program or other lifestyle management programs.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the MOVE! Program between 2006-2015 with attendance in at least 75% of classes for group A cohort.
* Completion of the MOVE! Program from 2012-2015 with participation in >75% of activities for group B cohort.
* The patient understands and has signed the study informed consent form.
* Veteran enrolled in the VA Healthcare System and followed by a VA primary care provider.

Exclusion Criteria:

* History of, or current diagnosed DSM-IV-TR eating disorder (i.e., anorexia nervosa or bulimia nervosa) or any current compensatory behaviors (e.g., vomiting, laxative use, excessive exercise).
* Individuals with prescription medication usage, or other medical/psychological conditions that could interfere with the physician's ability to assess the effect of the test results on weight loss.
* History of bipolar disorder, or organic brain syndromes; report hospitalization for any psychiatric disorder within the last 12 months.
* Are currently participating in a weight loss program and/or taking weight loss medication.
* Lost > 5% of body weight during the past 6 months or history of bariatric surgery.
* Failure to complete screening appointments.
* Health problems which may influence the ability to walk for physical activity or be associated with unintentional weight change, including cancer treatment within the past 5 years or tuberculosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US Veterans who have completed the MOVE! or TeleMOVE! program between 2011-2016
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Genetic SNP results | 3 months after start of MOVE! or TeleMOVE!
  Checking to see if our case control have different genotypes

REFERENCES:
- [Background] Ford ES, Giles WH, Dietz WH. Prevalence of the metabolic syndrome among US adults: findings from the third National Health and Nutrition Examination Survey. JAMA. 2002 Jan 16;287(3):356-9. doi: 10.1001/jama.287.3.356. PMID 11790215
- [Background] Ford ES, Li C, Sattar N. Metabolic syndrome and incident diabetes: current state of the evidence. Diabetes Care. 2008 Sep;31(9):1898-904. doi: 10.2337/dc08-0423. Epub 2008 Jun 30. PMID 18591398
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Koepsell TD, Littman AJ, Forsberg CW. Obesity, overweight, and their life course trajectories in veterans and non-veterans. Obesity (Silver Spring). 2012 Feb;20(2):434-9. doi: 10.1038/oby.2011.2. Epub 2011 Feb 3. PMID 21293452
- [Background] Kinsinger LS, Jones KR, Kahwati L, Harvey R, Burdick M, Zele V, Yevich SJ. Design and dissemination of the MOVE! Weight-Management Program for Veterans. Prev Chronic Dis. 2009 Jul;6(3):A98. Epub 2009 Jun 15. PMID 19527600
- [Background] Kahwati LC, Lance TX, Jones KR, Kinsinger LS. RE-AIM evaluation of the Veterans Health Administration's MOVE! Weight Management Program. Transl Behav Med. 2011 Dec;1(4):551-60. doi: 10.1007/s13142-011-0077-4. PMID 24073079